CLINICAL TRIAL: NCT00788177
Title: Subretinal Macugen® for Neovascular Age-Related Macular Degeneration (SUMANA)
Brief Title: Subretinal Macugen® for Neovascular Age-Related Macular Degeneration
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Klinikum Ludwigshafen (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Lars-Olof Hattenbach, MD, Privatdozent, Department of ophthalmology, Ludwigshafen hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AU-06102G
Record Dates: First submitted 2008-11-07; First posted 2008-11-10 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2009-07

CONDITIONS: Age-related Macular Degeneration
Keywords: age-related macular degeneration; subretinal injection; Pegaptanib; Macugen
MeSH Terms: conditions — Macular Degeneration | interventions — pegaptanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Pegaptanib (Macugen®) — Pegaptanib administered to the subretinal space (first dose) and to the vitreous cavity (following doses)
  Other Names: Macugen®, Pfizer Pharma GmbH

SUMMARY:
The purpose of this study is to assess the efficacy of pegaptanib (Macugen®) for neovascular (exudative) age-related macular degeneration (AMD) when the first dose is administered to the submacular space instead of vitreous body in cases when previous state-of-the-art treatment for the AMD was deemed ineffective.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 50 years and older with neovascular AMD proven by FA
* Patients who at baseline
* Have a BCVA letter score in the study eye between 20/40 to 20/320 using an ETDRS chart measured at 4 meters or Snellen equivalent
* Have a CNV lesion of any type in the study eye with the following characteristics as determined by fluorescein angiography:
* Evidence that CNV extends under the geometric center of the foveal avascular zone.
* Previous state-of-the-art therapy for the disease is deemed ineffective with following characteristics are given:
* Loss of visual acuity (2 or more Snellen lines) in the previous 3 months defined as either OR
* ≥10% increase in the lesion diameter as assessed by fluorescein angiography in the previous 3 months
* Ability of subject to understand character and individual consequences of clinical trial.
* Signed and dated informed consent of the subject must be available before start of any specific trial procedures.
* Women with childbearing potential practicing a medically accepted contraception (negative pregnancy test result, serum or urine at trial entry).

Exclusion Criteria:

* Subjects presenting with any of the following criteria will not be included in the trial:

  * Have a relevant ocular disease which may be associated with increased intraocular VEGF levels (namely uveitis, neovascular glaucoma, diabetic retinopathy, diabetic maculopathy, ocular ischemic syndrome, retinal vessel occlusion)
  * Had previous vitrectomy surgery for whatsoever reason
  * Are not pseudophakic
  * Have a >50% area of scarring of the whole CNV lesion size as seen in FA
  * Arterial hypertension refractory to medical treatment
  * Pregnancy and lactation.
  * History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product.
  * Participation in other clinical trials during the present clinical trial or within the last 3 months.
  * Medical or psychological condition that would not permit completion of the trial or signing of informed consent.
  * Suspected or present ocular or periocular infection

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-11; Primary Completion 2012-03 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who had lost fewer than 15 letters of visual acuity at 54 weeks | 54 weeks
Mean change from baseline in total size of lesion and total size of CNV at 12, 24 and 54 weeks | week 24 and 54

SECONDARY OUTCOMES:
Changes in best corrected visual acuity (BCVA) from baseline at 54 weeks | 54 weeks
Mean change from baseline in at week 12 and 24 | week 12 and 24
Proportion of patients who gain ≥ 5, 10, 15 letters of BCVA from baseline at week 24 and 54 | week 24 and 54
Proportion of patients who lose less than 15 letters of BCVA from baseline at week 24 and 54 | week 24 and 54
Change in area of leakage at 12, 24 and 54 weeks | weeks 12, 24 and 54
Mean change in retinal thickness by OCT at center of fovea at 12, 24 and 54 weeks | weeks 12, 24 and 54

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Olof Hattenbach, MD, Principal Investigator — Department of ophthalmology, Ludwigshafen hospital
Locations (1):
- Department of Ophthalmology, Ludwigshafen hospital, Ludwigshafen, Germany